CLINICAL TRIAL: NCT06684041
Title: Safety, Tolerability, Pharmacokinetic/Pharmacodynamic Study of Multiple Doses of HRS-5965 Capsules in Healthy Subjects and a Phase I Clinical Trial of the Effect of HRS-5965 on QT Interval in Healthy Subjects
Brief Title: A Safety, Tolerability, Pharmacokinetic/Pharmacodynamic Study, and QT Interval Study of HRS-5965 Capsules in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-5965-106
Record Dates: First submitted 2024-11-01; First posted 2024-11-12 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Hemolytic Anemia
MeSH Terms: conditions — Anemia, Hemolytic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose 1 (Experimental)
  Interventions: Drug: HRS-5965 capsule; Drug: HRS-5965 capsule placebo
- Dose 2 (Experimental)
  Interventions: Drug: HRS-5965 capsule; Drug: HRS-5965 capsule placebo
- Dose 3 (Experimental)
  Interventions: Drug: HRS-5965 capsule; Drug: HRS-5965 capsule placebo

INTERVENTIONS:
Drug: HRS-5965 capsule — HRS-5965 capsule
Drug: HRS-5965 capsule placebo — HRS-5965 capsule placebo

SUMMARY:
This was a randomized, double-blind, single-dose, placebo-controlled phase I clinical trial. This study plans to conduct three dose groups of dose 1, dose 2, and dose 3. A total of 32 healthy subjects were planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form before any activities related to this trial, be able to understand the procedures and methods of this trial, and be willing to complete this trial in strict accordance with the clinical trial protocol.
2. Aged between 18 and 45 years old (based on the time of signing the informed consent form), both males and females are eligible.
3. The body weight of males ≥ 50 kg, and that of females ≥ 45 kg, and body mass index (BMI): 19 - 26 kg/m².
4. During the screening period, there are no abnormalities in physical examination, vital signs, twelve - lead electrocardiogram, frontal and lateral chest radiographs, abdominal ultrasound, and laboratory tests, or those with minor abnormalities but judged by the investigator to be of no clinical significance.
5. During the screening period, human immunodeficiency virus antibody (HIV - Ab), treponema pallidum antibody, hepatitis B surface antigen (HBsAg), and hepatitis C virus antibody (HCV - Ab) are all negative.
6. Complete the vaccination of Neisseria meningitidis and Streptococcus pneumoniae vaccines 2 weeks before the first administration of HRS - 5965.

Exclusion Criteria:

1. The researcher has determined that there may be diseases or medical conditions that affect the absorption, distribution, metabolism and excretion of drugs or reduce compliance.
2. According to the judgment of the researcher, any physiological or psychological disease or condition that may increase the risk of the test, affect the subject's compliance with the protocol, or affect the subject's completion of the test.
3. Those with a previous history of Neisseria meningitidis infection, or those whose first - degree relatives have a history of Neisseria meningitidis infection.
4. Those with definite evidence of infection within 2 weeks before screening (positive etiological examination, or having received systemic antibiotic treatment), or those who have had a body temperature exceeding 38 °C.
5. Subjects with abnormal serum electrolytes (hypokalemia, hypomagnesemia, hypocalcemia).
6. Subjects with a history of convulsive disorders, long QT syndrome (including family history), syncope while swimming or any other type of syncope or history of loss of consciousness.
7. Subjects with a previous history of heart disease, such as hypertension, atherosclerosis, heart failure, bradycardia or stroke, or those using a pacemaker.
8. Those with a serum creatinine level exceeding the upper limit of the normal value, or those whose level does not exceed the upper limit but are judged by the investigator to be at risk of renal function impairment.
9. Those with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) exceeding the upper limit of normal value (ULN), or with total bilirubin exceeding 1.5 times the ULN.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-11-09 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Incidence of subjects with adverse events (AEs) | Baseline up to seven days after the last dosing.
  Incidence of AEs, including any abnormal findings in vital signs, and/or physical examination and/or clinical laboratory assessments and/or 12-lead ECG evaluation.
QTcF: Baseline and placebo-adjusted QTcF after oral HRS-5965 capsules | Baseline up to 24 hours after dosing.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to the time of last quantifiable analyte concentration (AUC0-t) for HRS-5965 | Baseline up to seven days after the last dosing.
Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-∞) for HRS-5965 | Baseline up to seven days after the last dosing.
Maximum plasma concentration (Cmax) for HRS-5965 | Baseline up to seven days after the last dosing.
Time to reach maximum plasma concentration (Tmax) for HRS-5965 | Baseline up to seven days after the last dosing.
Terminal half-life (t1/2) for HRS-5965 | Baseline up to seven days after the last dosing.
Apparent clearance (CL/F) of HRS-5965 for administration subcutaneously | Baseline up to seven days after the last dosing.
Apparent volume of distribution (V/F) of HRS-5965 for administration subcutaneously | Baseline up to seven days after the last dosing.
Complement system alternative pathway (AP) inhibition efficiency | Baseline up to seven days after the last dosing.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided